CLINICAL TRIAL: NCT01599442
Title: Register for Patients With Diabetic Foot Syndrome and Critical Limb Ischemia
Acronym: August-1
Status: Terminated | Type: Observational
Why Stopped: recrution number was not reached
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: August-1
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Foot; Critical Limb Ischemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diabetic foot syndrome (DFS) is a disease caused by neurogenic (concerning the nervous system), vascular, mechanic and metabolic factors, which are further complicated by an impairment of the immune system and a corresponding increase in the risk for infections. Results from clinical trials about the efficacy of interventions aimed at reducing the number of patient-relevant end points are of limited comparability due to the heterogenity of patient characteristics. By their very nature, randomized clinical trials (RCT) can only focus on a limited section of the wide range of possible intervention regimes. In clinical practice, however, a number of patients with dfs will never have been part of a clinical trial. Furthermore, there are only very few contemporary registers for this indication from which conclusions with regard to the comparative merits of different therapeutic strategies may be drawn.

The register was conceived to find out to which extent RCT patients are representative for the overall patient collective with dfs and critical limb ischemia and to evaluate the therapeutic success of other treatment strategies. An RCT to assess the efficacy of urokinase versus placebo is imbedded in the register.

DETAILED DESCRIPTION:
August-1 is a register to find out to which extent RCT patients are representative for the overall patient collective with dfs and critical limb ischemia and to evaluate the therapeutic success of other treatment strategies. An RCT to assess the efficacy of urokinase versus placebo is imbedded in the register.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with dfs and critical limb ischemia
* age 18 and older

Exclusion Criteria:

* less than 1 year life expectancy
* prior major amputation
* planned major expectation
* prior treatment of the current episode of dfs with urokinase
* mechanical heart valve replacement
* cerebral event with changes in CT during the last three months
* non-remediated proliferating retinopathy
* uncontrolled hypertension (systolic > 180 mmHg, diastolic > 100 mmHg)
* hemorrhagic diathesis (spontaneous quick value < 50%, spontaneous ptt > 40 sec, thrombocytes < 100 gpt/l)
* acute gastrointestinal bleeding or ulcers during the last 4 weeks
* prior reverse bypass operation
* concomitant participation in other clinical trials
* insufficient compliance
* premenopausal women not using a safe method of contraception (i. e. IUD, hormone implants, hormone depot injection, combined pill (estrogens and gestagens), vaginal ring or vasectomized partner).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients from hospitals with a department specializing in the treatment of diabetic foot syndrome
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
duration of survival without major amputation | to be assessed after 12 months observation

SECONDARY OUTCOMES:
major amputation | after 12 months observation
total mortality | after 12 months observation

CONTACTS AND LOCATIONS:
Overall Officials: S. Schellong, Prof.Dr.med., Principal Investigator — Staedt. KH Dresden-Friedrichstadt
Locations (1):
- Krankenhaus Dresden-Friedrichstadt, Dresden, Sachse, Germany